CLINICAL TRIAL: NCT00955734
Title: Early Motion After Volar Fixation for Distal Radius Fractures: A Prospective Trial
Brief Title: Early Motion After Volar Fixation for Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ryan Calfee, MD, Associate Professor of Orthopaedic Surgery, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-0566
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Radius Fracture
Keywords: wrist; fracture; motion; surgery
MeSH Terms: conditions — Radius Fractures; Fractures, Bone | interventions — Immobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early motion (Experimental): This group of patients will begin wrist motion 1 week after surgery.
  Interventions: Other: Early motion
- Immobilization (Active Comparator): This group will be casted for 6 weeks after surgery
  Interventions: Other: Immobilization

INTERVENTIONS:
Other: Early motion — One set of patients will begin wrist motion at 1 week after surgery.
  Arms: Early motion
Other: Immobilization — This set of patients will be casted for 6 weeks after surgery.
  Arms: Immobilization

SUMMARY:
Many surgeons pursue volar plating of the distal radius to allow earlier post-operative wrist motion. Early motion is generally prescribed in the belief that it will result in greater final motion without compromising fixation. However, studies have failed to demonstrate clinically significant improvement in final wrist motion (> 1 year follow up) compared to treatments requiring longer immobilization such as external fixation or bridge plating.

DETAILED DESCRIPTION:
Many surgeons pursue volar plating of the distal radius to allow earlier post-operative wrist motion. Early motion is generally prescribed in the belief that it will result in greater final motion without compromising fixation. However, studies have failed to demonstrate clinically significant improvement in final wrist motion (>1 year follow up) compared to treatments requiring longer immobilization such as external fixation or bridge plating (McQueen 1996, Handoll 2003, Atroshi 2006, Krishnan 2003, Sommerkamp 1994, Grewal 2005).

Only one study to date has attempted to define the early effects of wrist mobilization following volar plate fixation of the distal radius (Lozano-Calderon 2008). That study prospectively enrolled 60 patients and randomized them to begin wrist motion at 2 weeks (range 7 days - 13 days) or 6 weeks (range 42 to 49 days) postoperatively. This study found no significant difference in subjective or objective outcome measures at 3 or 6 months follow up. However, the investigation had several weaknesses. First, there was no attempt to confirm adherence to the immobilization protocols. Those in the late motion group were not casted but remained in orthoplast splints which could be easily removed. Secondly, this investigation collected data only at 3 and 6 months which prohibited them from commenting on the rate of improvement during the early weeks after mobilization. The authors acknowledged these limitations and further noted that no evaluation of patient cost was performed. Finally, radiographic evaluations in this study did not include analysis of change in alignment from immediate postoperative films.

Thus, the literature to date suggests that early mobilization of the volarly plated distal radius is safe but does not improve final wrist motion. The benefits of mobilization in the early postoperative period though have not been clearly defined. This project proposes to fill this void in the literature and determine if early mobilization is an effective measure to hasten recovery of motion and function.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age having volar internal fixation for distal radius fractures.

Exclusion Criteria:

* Patients will be excluded if immobilization is required for distal radioulnar joint instability (whether operatively pinned or simply immobilized in supination) or an associated carpal injury.
* Patients with concurrent fracture of the ulna proximal to the base of the ulnar styloid will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Wrist Motion | 2 weeks - 1 year

SECONDARY OUTCOMES:
Patient Function | 2 weeks - 1 year
Patient Pain | 2 weeks - 1 year
Fracture reduction | 2 week - 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Calfee, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States